CLINICAL TRIAL: NCT02324621
Title: A Continuation Clinical Trial of Every Three-Week Dosing of Oral ONC201 in Patients With Advanced Solid Tumors
Brief Title: Continuation of Oral ONC201 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other); Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 051407; NCI-2014-02043 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 051407 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-12-24 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Unspecified Adult Solid Tumor
Keywords: protocol specific
MeSH Terms: interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (oral ONC201) (Experimental): Patients receive oral ONC201 PO on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oral ONC201; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Oral ONC201 — Given PO
  Other Names: ONC201; TIC10
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the long-term side effects of the continuation of oral ONC201 in treating patients with solid tumors that have spread to other places in the body who have previously benefited from receiving this drug. Oral ONC201 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the long-term safety and tolerability of ONC201 (oral ONC201) administered orally in patients with advanced cancers.

SECONDARY OBJECTIVES:

I. To characterize pharmacokinetics of ONC201. II. To assess serum biomarkers of therapeutic response to ONC201. III. To assess preliminary antitumor activity of ONC201 as a single agent in advanced solid tumors.

OUTLINE:

Patients receive oral ONC201 orally (PO) on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed participation in one of the ONC201 protocols, has not shown tumor progression while on study treatment, and has tolerated the study drug without unacceptable toxicities
* Patient has not met criteria for withdrawal from the base protocol
* Patient is willing to comply with protocol requirements and procedures, and keep scheduled study visits
* Patient agrees to practice effective contraception during the entire study period unless documentation of infertility exists
* Patient is able to understand and is willing to sign the informed consent form

Exclusion Criteria:

* Patient is receiving concomitant standard and/or investigational anticancer therapy; local palliative radiotherapy is permissible upon discussion with the principal investigator
* Patient has alcohol or substance abuse which, in the opinion of the investigator, would interfere with compliance or safety
* Patient has any condition or laboratory abnormality which, in the opinion of the investigator, would pose additional risk in administering the study drug to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse experiences from oral ONC201 using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 4 weeks after end of study treatment
  An adverse experience is defined as any unintended or abnormal clinical observation that is not of benefit to the patient. Either the condition was not present prior to exposure to the study therapy, or it has worsened in intensity or frequency following exposure to the study therapy. Descriptive statistics will be provided.

SECONDARY OUTCOMES:
Frequency of toxicities associated with ONC201 | Up to 4 weeks after end of study treatment
Response rate of oral ONC201 in patients with advanced solid tumors | At 3 months
Pharmacokinetic parameters | Up to 4 weeks of therapy
  The oral ONC201 concentration, and the corresponding time, area under the curve, elimination half-life, total body clearance and volume of distribution will be determined for each patient concentration-time data using a non-compartmental model. Descriptive statistics will be provided.
Clinical benefit rate (stable disease and partial disease) | At 3 months
Time to progressive disease | Up to 4 weeks after end of study treatment
  Descriptive statistics on continuous data will include means, medians, standard deviations, and ranges will be provided to estimate clinical benefit rate.

OTHER OUTCOMES:
Changes in serum biomarkers of therapeutic response | Baseline to up to 4 weeks after end of study treatment
  Descriptive statistics will be provided.
Changes in molecular targets of oral ONC201 | Baseline to up to 4 weeks after end of study treatment
  Descriptive statistics will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Malhotra, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Stein MN, Malhotra J, Tarapore RS, Malhotra U, Silk AW, Chan N, Rodriguez L, Aisner J, Aiken RD, Mayer T, Haffty BG, Newman JH, Aspromonte SM, Bommareddy PK, Estupinian R, Chesson CB, Sadimin ET, Li S, Medina DJ, Saunders T, Frankel M, Kareddula A, Damare S, Wesolowsky E, Gabel C, El-Deiry WS, Prabhu VV, Allen JE, Stogniew M, Oster W, Bertino JR, Libutti SK, Mehnert JM, Zloza A. Safety and enhanced immunostimulatory activity of the DRD2 antagonist ONC201 in advanced solid tumor patients with weekly oral administration. J Immunother Cancer. 2019 May 22;7(1):136. doi: 10.1186/s40425-019-0599-8. PMID 31118108